CLINICAL TRIAL: NCT03549260
Title: Randomized, Double-Blind, Placebo-Controlled, Phase 2, Dose Finding Study to Evaluate the Efficacy and Safety of LIB003 in Patients on Stable Lipid-Lowering Therapy Requiring Additional LDL-C Reduction
Brief Title: Study to Evaluate Efficacy and Safety of LIB003 in Patients on Lipid-Lowering Therapy Needing Additional LDL-C Reduction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LIB Therapeutics LLC (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIB003-002
Record Dates: First submitted 2018-05-22; First posted 2018-06-07 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: LDL Cholesterol
Keywords: low density lipoprotein cholesterol; PCSK9

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled trial to evaluate LDL-C reduction with 3 different doses of LIB003 compared to placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind and Placebo-Controlled - Study drug administered by unmasked nurse who is not involved in any other aspects of the trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LIB003 150 mg or matching placebo (Experimental): SC LIB003 150 mg or placebo every 4 weeks
  Interventions: Biological: LIB003
- LIB003 300 mg or matching placebo (Experimental): SC LIB003 300 mg or placebo every 4 weeks
  Interventions: Biological: LIB003
- LIB003 350 mg or matching placebo (Experimental): SC LIB003 350 mg or placebo every 4 weeks
  Interventions: Biological: LIB003

INTERVENTIONS:
Biological: LIB003 — LIB003 or placebo

SUMMARY:
Study to assess the LDL-C lowering efficacy of different doses of LIB003 administered every 4 weeks in subjects on stable statin and/or ezetimibe therapy

DETAILED DESCRIPTION:
Randomized, Double-Blind, Placebo-Controlled, Phase 2 study to assess the LDL-C lowering efficacy at Week 12 of various doses of LIB003 administered subcutaneously (SC) every 4 weeks (Q4W) in patients with hypercholesterolemia on stable diet and oral LDL-C-lowering drug therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older
2. Elevated LDL-C on current lipid lowering therapy and; prior atherosclerotic cardiovascular disease (ASCVD) event or evidence of ASCVD or without ASCVD but at high risk for ASCVD based on AHA/ACC CVD risk calculator, or aged 40 years and older with diabetes and moderate- to high-intensity statin, or pre-treatment LDL-C 190 mg/dL or greater or heterozygous familial hypercholesterolemia (HeFH)
3. Body mass index (BMI) between 18 and 40 kg/m2

Exclusion Criteria:

1. Females of childbearing potential not using or willing to use an effective form of contraception, or pregnant or breastfeeding, or who have a positive serum pregnancy test at screening
2. Homozygous familial hypercholesterolemia
3. LDL or plasma apheresis within 2 months; lomitapide or mipomersen within 12 months
4. Uncontrolled cardiac arrhythmia, myocardial infarction, unstable angina, PCI, CABG, or stroke within 3 months prior to enrollment
5. Uncontrolled cardiac arrhythmia, myocardial infarction, unstable angina, PCI, CABG, or stroke within 3 months prior to enrollment
6. Newly diagnosed or poorly controlled (HbA1c >9%) type 2 diabetes
7. Uncontrolled hypertension
8. Moderate to severe renal insufficiency
9. Elevated liver function test at screening
10. Uncontrolled cardiac arrhythmia or prolonged QT on EKG
11. A history of prescription drug abuse, illicit drug use, or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Percent reduction in Low Density Lipoprotein Cholesterol (LDL-C) at week 12 | baseline to 12 weeks
  Change in serum LDL-C from baseline after 12 weeks

SECONDARY OUTCOMES:
The incidence and severity of treatment emergent adverse events (TEAEs) | baseline to 12 weeks
  safety and tolerability will be based on the incidence and severity of treatment emergent adverse events
Percent reduction in apolipoprotein B (Apo B) at week 12 | baseline to 12 weeks
  Change in serum Apo B from baseline after 12 weeks
Percent reduction in lipoprotein (a) [Lp(a)] at week 12 | baseline to 12 weeks
  Change in serum Lp(a) from baseline after 12 weeks
Percent reduction in free PCSK9 at week 12 | baseline to 12 weeks
  Change in serum free PCSK9 from baseline after 12 weeks
Presence of anti LIB003 antibodies (ADAs) | baseline to 12 weeks
  Measurement of ADAs at baseline and various intervals

CONTACTS AND LOCATIONS:
Overall Officials: Evan A Stein, MD, Study Director — LIB Therapeutics LLC
Locations (5):
- United States (5):
  - Midwest Institute For Clinical Research, Indianapolis, Indiana
  - Louisville Metabolic and Atherosclerosis Research Center, Louisville, Kentucky
  - Sterling Research Group, Cincinnati, Ohio
  - The Lindner Research Center, Cincinnati, Ohio
  - Metabolic & Atherosclerosis Research Center (MARC), Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Informed Consent Form (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT03549260/ICF_001.pdf
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT03549260/Prot_002.pdf